CLINICAL TRIAL: NCT04860271
Title: Comparison of Manual Acupuncture Effectivity Using Filiform Needles and Press Tack Needle for Healthcare Worker's Anxiety During COVID-19 Outbreak: A Randomized Clinical Trial
Brief Title: Manual Acupuncture Using Acupuncture Needle vs Press Needle for COVID-19 Healthcare Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. Irma Nareswari, B.MedSc, Sp.Ak, Head of Medical Acupuncture Study Programme University of Indonesia, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-12-1513
Record Dates: First submitted 2021-04-23; First posted 2021-04-26 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Anxiety
Keywords: acupuncture; press needle; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator did not know the respondent and did not come in contact. The outcome assessor consist of 4 person who are randomly assessing the respondent, so the assessor do not know the full data since the beginning of participation thus do not have any bias when assessing the respondent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Filiform Needle (Active Comparator): Respondent are health workers that is having mild to moderate anxiety symptoms, with Hamilton Anxiety Scale less than 25. This arm will receive 6 acupuncture treatment within 2 weeks, and will be taken outcome measurements 4 times, that is before the first treatment, after the third treatment, after the sixth treatment and at 2 weeks after the sixth treatment.
  Interventions: Procedure: Manual Acupuncture
- Press Needle (Active Comparator): Respondent are health workers that is having mild to moderate anxiety symptoms, with Hamilton Anxiety Scale less than 25. This arm will receive 3 acupuncture treatment within 2 weeks, and will be taken outcome measurements 4 times, that is before the first needle placement, after replacing the first sets of needles, after removing the third sets of needles and at 2 weeks after removing the third sets of needle.
  Interventions: Procedure: Manual Acupuncture

INTERVENTIONS:
Procedure: Manual Acupuncture — Manual acupuncture treatment using different types of needle

SUMMARY:
This study would like to compare manual acupunture treatment for anxiety in COVID Health workers population in Cipto Mangunkusumo Hospital using filiform needles and press needle.

DETAILED DESCRIPTION:
This study wanted to know would press needle be having better outcome for anxiety treatment, compared with filiform needles, because press needle taken home and could be manipulated as needed at home, unlike filiform needle where an acupuncturist must be available to do the treatment. Furthermore, the press needle needed to be changed once within 5 days, that is 2-3 times in week. So we hope to have better acupuncture option (in effectivity and timewise) for COVID healthcare workers anxiety treatment. There are no study to compare the usage of the two types of needles for anxiety treatment to date.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 health workers.
* Rapid test COVID-19 t or PCR swab non reactive within 7 days before intervention
* HAM-A score below 25
* Could still do daily activities
* Willing to enroll this study and sign the informed consent
* Willing to comply with the study procedure

Exclusion Criteria:

* Contraindicated for acupuncture : having medical emergencies, pregnancy, blood clotting issue, uncontrolled diabetic mellitus, fever.
* Having acupunture treatment within 7 days prior to study intervention
* Having tumor or infection at the pucture site
* Cognitive or consciouseness impairment
* Having anxiety therapy with a psychiatrist

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale | two weeks
  A questionnaire to access anxiety level, higher score means higher anxiety symptoms, ranged 0-56, mild anxiety scored below 17, 17-24 moderate anxiety, more than 24 severe anxiety
Short-Form 36 | two weeks
  A questionnaire to access quality of life, higher score means better quality of life. ranged 1-100. higher scores means better quality of life

SECONDARY OUTCOMES:
Heart Rate Variability | two weeks
  A measurement to know the balance of autonomic nerve system

CONTACTS AND LOCATIONS:
Overall Officials: Irma Nareswari, dr. Sp.Ak, Principal Investigator — Faculty of Medicine, University of Indonesia
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: No